CLINICAL TRIAL: NCT01854151
Title: Promoting Safe Use of Pediatric Liquid Medications: A Health Literacy Approach
Brief Title: Promoting Safe Use of Pediatric Liquid Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Emory University (Other); Northwestern University (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-01122; 1R01HD070864-01A1 (NIH)
Record Dates: First submitted 2013-05-14; First posted 2013-05-15 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Medication Errors
Keywords: Medication errors; Medication dosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Practice (No Intervention): Parents whose children are prescribed medication and meet inclusion/exclusion criteria will fill their medication at their regular pharmacy and receive medication with labeling and dosing instruments as per routine
- New Labeling/Dosing Strategy (Experimental): Parents whose children are prescribed liquid medication and meet inclusion/exclusion criteria will receive medications with health literacy informed labels and dosing instruments
  Interventions: Other: New Labeling/Dosing Strategy

INTERVENTIONS:
Other: New Labeling/Dosing Strategy — Parents whose children are prescribed liquid medication will receive medications with health literacy informed labels and dosing instruments
  Arms: New Labeling/Dosing Strategy

SUMMARY:
Variable and poor-quality drug labeling has been cited as a leading cause of medication errors and adverse drug events, especially in the context of low health literacy. This is a particularly important issue in pediatrics as more than half of US children are exposed to one or more outpatient medications in a given week, and studies suggest that over half of caregivers make errors when dosing liquid medications for children. Our study objective is to identify evidence-based strategies for labeling and dosing prescription and over-the-counter pediatric liquid medications in order to promote safe, appropriate use, as well as to inform state and federal policy standards. We hypothesize that a health literacy-informed labeling and dosing strategy will result in improved parent ability to administer medications prescribed to their young children.

DETAILED DESCRIPTION:
Administering pediatric medications is frequently a difficult task for parents, in large part due to reliance on liquid formulations requiring the use of confusing, and often complex, measurement devices. Use of different units of measurement (milliliter, teaspoon, and/or tablespoon units) with variations in associated abbreviations, and the variability of measuring devices (type, markings, capacity), are sources of parent confusion. Low health literacy is linked to caregiver misunderstanding. Despite high error and utilization rates for outpatient pediatric medications, research examining strategies to prevent medication errors have focused largely on adults and on inpatient populations.

The ability to understand pediatric medication instructions is a critical health literacy and patient safety concern. Recently, the US Food and Drug Administration recognized the importance of this issue and released new guidelines to promote improved labeling and measuring devices for pediatric liquid medications. While these recommendations are an essential first step, evidence is needed to support the development of 'best practices' for designing optimal instructions and devices, especially for parents with limited literacy and/or limited English proficiency.

Our study objective is to identify evidence-based 'best practices' for labeling and dosing prescription and over-the-counter pediatric liquid medications in order to promote safe, appropriate use. A series of experiments will first be conducted to examine the efficacy of specific dosing and measurement strategies for improving parent understanding and use of pediatric liquid medications, including examining the impact of milliliter-only label instructions and devices, as well as the potential role for pictographic dosing diagrams. Findings will be merged with existing evidence-based health literacy 'best practices' for medication labeling to develop a comprehensive, patient-centered strategy for the labeling and dosing of pediatric liquid medications. The effectiveness of the patient-centered strategy will then be evaluated as part of a randomized controlled trial among English and Spanish-speaking parents whose children have been newly prescribed oral liquid antibiotics in a pediatric emergency department setting. Secondary aims of the study include extending the body of literature on health literacy and pediatric medication use, and generating a policy road map for achieving and implementing labeling and dosing standards for pediatric liquid medications.

ELIGIBILITY:
Phase II of Study (Effectiveness Trial)

Inclusion Criteria:

* parent/legal guardian of a child age 8 or less
* parent/legal guardian age 18 or greater
* child presenting for care in the emergency department
* child prescribed short course liquid antibiotic
* parent English or Spanish-speaking
* parent responsible for administering medication to child

Exclusion Criteria:

* parent visual acuity worse than 20/50 (Rosenbaum Pocket Screener)
* parent with uncorrectable hearing impairment
* prior participation in study involving medication dosing

Max Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1005 (Actual)
Dates: Start 2013-04-22 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Medication dosing accuracy | Target within 2 weeks after medication course completion

CONTACTS AND LOCATIONS:
Overall Officials: H. Shonna Yin, MD, MS, Principal Investigator — NYU School of Medicine / Bellevue Hospital Center
Locations (4):
- United States (4):
  - Stanford University School of Medicine, Stanford, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - New York University School of Medicine, New York, New York

REFERENCES:
- [Derived] Yin HS, Parker RM, Sanders LM, Dreyer BP, Mendelsohn AL, Bailey S, Patel DA, Jimenez JJ, Kim KA, Jacobson K, Hedlund L, Smith MC, Maness Harris L, McFadden T, Wolf MS. Liquid Medication Errors and Dosing Tools: A Randomized Controlled Experiment. Pediatrics. 2016 Oct;138(4):e20160357. doi: 10.1542/peds.2016-0357. Epub 2016 Sep 12. PMID 27621414